CLINICAL TRIAL: NCT05783414
Title: Effectiveness and Cost-effectiveness of Virtually Delivered Cognitive Stimulation Therapy (vCST) and Online Dementia Carer Support
Brief Title: Effectiveness and Cost-effectiveness of vCST and Online Dementia Carer Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: City University of Hong Kong (Other); University of Auckland, New Zealand (Other); London School of Economics and Political Science (Other); Chinese University of Hong Kong (Other); University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: C7055-21GF
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Dementia
Keywords: cognitive stimulation therapy (CST); virtually delivered cognitive stimulation therapy (vCST); carer support programme; information and communication technology (ICT); cluster randomised trial; effectiveness; cost-effectiveness; Chinese
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The researchers performing the assessments will be blinded to the intervention group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- vCST + f2f carer support (Experimental): vCST followed by in-person carer support programme
  Interventions: Behavioral: f2f carer support; Behavioral: vCST
- f2f CST + f2f carer support (Active Comparator): In-person CST followed by in-person carer support programme
  Interventions: Behavioral: f2f CST; Behavioral: f2f carer support
- vCST + online carer support (Experimental): vCST followed by online carer support programme
  Interventions: Behavioral: vCST; Behavioral: online carer support
- f2f CST + online carer support (Experimental): In-person CST followed by online carer support programme
  Interventions: Behavioral: f2f CST; Behavioral: online carer support

INTERVENTIONS:
Behavioral: f2f CST — An evidence-based group CST protocol adapted for Hong Kong Chinese culture. It consists of 14 sessions of group activities (group size: 6) for people with mild to moderate dementia, where participants with similar level of cognitive impairment receive cognitively stimulating social activities twice per week over 7 weeks.
  Arms: f2f CST + f2f carer support; f2f CST + online carer support
Behavioral: f2f carer support — Centre-based carer support programme for dementia carers provided in a community care service centre, which provide group education on caring skills, mutual support groups, and group-based self-care training over 6 months.
  Arms: f2f CST + f2f carer support; vCST + f2f carer support
Behavioral: vCST — A home-based version of f2f CST delivered via an information and communication technology platform (Zoom plus a web-based CST platform). It consists of 14 sessions of group activities (group size: 3) for people with mild to moderate dementia, where participants with similar level of cognitive impairment receive cognitively stimulating social activities twice per week over 7 weeks.
  Arms: vCST + f2f carer support; vCST + online carer support
Behavioral: online carer support — A home-based carer support service delivered via an information and communication technology platform (Zoom plus a web-based carer platform). It consists of 4 group sessions (group size: 6) and 3 individual sessions, and 3 optional self-learning sessions over 6 months, with an empowering care management approach to strengthen carer self-efficacy.
  Arms: f2f CST + online carer support; vCST + online carer support

SUMMARY:
A multicentre single-blind cluster randomised trial to evaluate the effectiveness and cost-effectiveness of virtually delivered versus in-person cognitive stimulation therapy (CST) and carer support in people living with dementia and carers

DETAILED DESCRIPTION:
This is a multicentre, single-blind cluster randomised trial with an aim to evaluate the effectiveness and cost-effectiveness of virtual delivery of CST and carer support in comparison with in-person CST and carer support in Hong Kong Chinese. A total of 156 dyads of people living with dementia and carers will be randomly assigned to one of the four groups: (A) vCST (7 weeks) followed by in-person carer support programme (6 months); (B) in-person CST (7 weeks) followed by in-person carer support programme (6 months); (C) vCST (7 weeks) followed by online carer support programme (6 months); and (D) in-person CST (7 weeks) followed by online carer support programme (6 months). The investigators will measure outcomes at baseline, 7 weeks, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* having a clinical diagnosis of mild to moderate dementia;
* having a family carer;
* living in the community in Hong Kong;
* able to communicate and understand communication;
* able to see and hear well enough to participate in a meaningful assessment;
* the person with dementia and/or his/her carer can provide informed consent

Exclusion Criteria:

* unable to communicate;
* unable to participate in intervention due to significant hearing or visual impairment, or other physical or psychiatric conditions

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Change in cognitive function | From T0 (baseline) to T1 (7 weeks)
  Change in cognitive function in persons living with dementia measured using the Chinese version of the Alzheimer's Disease Assessment Scale - Cognitive section (ADAS-Cog) from T0 (baseline) to T1 (7 weeks).
Change in quality of life in persons living with dementia | From T0 (baseline) to T1 (7 weeks)
  Change in quality of life in persons living with dementia measured using the 13-item Quality of Life in Alzheimer's Disease (QoL-AD) from T0 (baseline) to T1 (7 weeks).
Change in self-efficacy | From T1 (7 weeks) to T2 (6 months post-CST)
  Change in self-efficacy in dementia carers measured using the Chinese Revised Scale for Caregiving Self-Efficacy (CSE-R) from T1 (7 weeks) to T2 (6 month post-CST).

SECONDARY OUTCOMES:
Change in behavioural and psychological symptoms of dementia | From T0 (baseline) to T2 (6 months post-CST)
  Change in behavioural and psychological symptoms of dementia measured using the Neuropsychological Inventory Questionnaire (NPI-Q), a 12-item informant-based interview from T0 (baseline) to T2 (6 months post-CST).
Change in functioning | From T0 (baseline) to T2 (6 months post-CST)
  Change in functioning of the persons living with dementia measured using the Chinese version of the Disability Assessment for Dementia (CDAD), an informant-based assessment, from T0 (baseline) to T2 (6 months post-CST).
Change in mental wellbeing (PLwD) | From T0 (baseline) to T1 (7 weeks)
  Change in mental wellbeing in the persons living with dementia measured using the Short Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS), which has been validated in Hong Kong and used in people living with dementia, from T0 (baseline) to T1 (7 weeks).
Change in carer burden | From T0 (baseline) to T2 (6 months post-CST)
  Change in carer burden measured using the Chinese 12-item version Zarit Burden Interview (CZBI) in carer from T0 (baseline) to T2 (6 months post-CST).
Change in mental wellbeing (carer) | From T0 (baseline) to T2 (6 months post-CST)
  Change in mental wellbeing in carers measured using the WEMWBS from T0 (baseline) to T2 (6 months).
Change in social functioning | From T0 (baseline) to T1 (7 weeks)
  Change in social functioning in the persons living with dementia measured using the Hong Kong version of Social Functioning in Dementia Scale (HKSF-DEM), a self-rating and proxy rating scale, from T0 (baseline) to T1 (7 weeks).
Change in health-related quality of life (PLwD) | From T0 (baseline) to T1 (7 weeks)
  Change in health-related quality of life in the persons living with dementia measured using the EQ-5D-5L, a self-rating and proxy-rating scale, from T0 (baseline) to T1 (7 weeks).
Change in perceived positive aspects of caregiving | From T1 (7 weeks) to T2 (6 months post-CST)
  Change in perceived positive aspect of caregiving in carers measured using the Positive Aspect of Caregiving Scale (PAC) from T1 (7 weeks) to T2 (6 months post-CST).
Change in health-related quality of life (carer) | From T0 (baseline) to T2 (6 months post-CST)
  Change in health-related quality of life in carers measured using the EQ-5D-5L, a self-rating and proxy-rating scale, from T0 (baseline) to T2 (6 months post-CST).

OTHER OUTCOMES:
Extent to meet and attain a set of pre-agreed goals | 6 months
  The Goal Attainment Scale (GAS) would be used to record a set of goals the carer desires to achieve in T1 (7 weeks) and assess the extent of goal achievement in T2 (6 months).
Types and level of engagement | 7 weeks
  An observational tool of engagement adapted from the Myers Research Institute Engagement Scale (MRI-ES) would be used to assess the types and level of engagement of persons living with dementia during CST intervention.
Change in spontaneous speech and discourse production | From T0 (baseline) to T1 (7 weeks)
  Change in spontaneous speech and discourse production in persons living with dementia assessed using short conversation, important event recall, and picture description from T0 (baseline) to T1 (7 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Wong, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prince M, Bryce R, Ferri C, Alzheimer's Disease International. World Alzheimer Report 2011: The Benefits of Early Diagnosis and Intervention. London, UK: Alzheimer's Disease International; 2011.
- [Background] Woods B, Aguirre E, Spector AE, Orrell M. Cognitive stimulation to improve cognitive functioning in people with dementia. Cochrane Database Syst Rev. 2012 Feb 15;(2):CD005562. doi: 10.1002/14651858.CD005562.pub2. PMID 22336813
- [Background] Knapp M, Thorgrimsen L, Patel A, Spector A, Hallam A, Woods B, Orrell M. Cognitive stimulation therapy for people with dementia: cost-effectiveness analysis. Br J Psychiatry. 2006 Jun;188:574-80. doi: 10.1192/bjp.bp.105.010561. PMID 16738349
- [Background] Dementia: Assessment, management and support for people living with dementia and their carers. London: National Institute for Health and Care Excellence (NICE); 2018 Jun. Available from http://www.ncbi.nlm.nih.gov/books/NBK513207/ PMID 30011160
- [Background] Dai R, Zhang AY, Wong G. The impact of covid19 on formal and informal dementia care in Hong Kong. 34th International Conference of Alzheimer's Disease International; 2020.
- [Background] Chu LW, Chiu KC, Hui SL, Yu GK, Tsui WJ, Lee PW. The reliability and validity of the Alzheimer's Disease Assessment Scale Cognitive Subscale (ADAS-Cog) among the elderly Chinese in Hong Kong. Ann Acad Med Singap. 2000 Jul;29(4):474-85. PMID 11056778
- [Background] Chan IW, Chu LW, Lee PW, Li SW, Yu KK. Effects of cognitive function and depressive mood on the quality of life in Chinese Alzheimer's disease patients in Hong Kong. Geriatr Gerontol Int. 2011 Jan;11(1):69-76. doi: 10.1111/j.1447-0594.2010.00643.x. Epub 2010 Aug 25. PMID 20738410
- [Background] Tang JY, Ho AH, Luo H, Wong GH, Lau BH, Lum TY, Cheung KS. Validating a Cantonese short version of the Zarit Burden Interview (CZBI-Short) for dementia caregivers. Aging Ment Health. 2016 Sep;20(9):996-1001. doi: 10.1080/13607863.2015.1047323. Epub 2015 May 27. PMID 26016419
- [Background] Sun Y, Luk TT, Wang MP, Shen C, Ho SY, Viswanath K, Chan SSC, Lam TH. The reliability and validity of the Chinese Short Warwick-Edinburgh Mental Well-being Scale in the general population of Hong Kong. Qual Life Res. 2019 Oct;28(10):2813-2820. doi: 10.1007/s11136-019-02218-5. Epub 2019 May 29. PMID 31144205
- [Background] Wong A, Cheng ST, Lo ES, Kwan PW, Law LS, Chan AY, Wong LK, Mok V. Validity and reliability of the neuropsychiatric inventory questionnaire version in patients with stroke or transient ischemic attack having cognitive impairment. J Geriatr Psychiatry Neurol. 2014 Dec;27(4):247-52. doi: 10.1177/0891988714532017. Epub 2014 Apr 24. PMID 24763069
- [Background] Au A, Lai MK, Lau KM, Pan PC, Lam L, Thompson L, Gallagher-Thompson D. Social support and well-being in dementia family caregivers: the mediating role of self-efficacy. Aging Ment Health. 2009 Sep;13(5):761-8. doi: 10.1080/13607860902918223. PMID 19882415
- [Background] Judge KS, Camp CJ, Orsulic-Jeras S. Use of Montessori-based activities for clients with dementia in adult day care: Effects on engagement. American Journal of Alzheimer's Disease 2000; 15(1): 42-6.
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Chisholm D, Knapp MR, Knudsen HC, Amaddeo F, Gaite L, van Wijngaarden B. Client Socio-Demographic and Service Receipt Inventory--European Version: development of an instrument for international research. EPSILON Study 5. European Psychiatric Services: Inputs Linked to Outcome Domains and Needs. Br J Psychiatry Suppl. 2000;(39):s28-33. doi: 10.1192/bjp.177.39.s28. PMID 10945075
- [Background] Lu S, Liu T, Wong GHY, Leung DKY, Sze LCY, Kwok WW, Knapp M, Lou VWQ, Tse S, Ng SM, Wong PWC, Tang JYM, Lum TYS. Health and social care service utilisation and associated expenditure among community-dwelling older adults with depressive symptoms. Epidemiol Psychiatr Sci. 2021 Feb 2;30:e10. doi: 10.1017/S2045796020001122. PMID 33526166